CLINICAL TRIAL: NCT01943188
Title: Pilot Study of Local Tumor Irradiation With Autologous T-Cell Infusion for Metastatic Renal Cell Carcinoma
Brief Title: Stereotactic Body Radiation Therapy and T-Cell Infusion in Treating Patients With Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sandy Srinivas, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RENAL0027; NCI-2013-01688 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RENAL0027 (Other: Stanford University Hospitals and Clinics); P30CA124435 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery; Cyclophosphamide

ARMS (1):
- Treatment (SBRT, autologous PBMC infusion) (Experimental): SBRT: Patients undergo standard of care SBRT over 1-2 weeks according to tumor volume and location.
  LYMPHODEPLETION: Beginning 3 weeks later, patients receive cyclophosphamide PO BID for 3 days.
  REINFUSION OF PBMC: Within 3-14 days of completing lymphodepletion with cyclophosphamide , patients undergo autologous PBMC infusion.
  Interventions: Radiation: stereotactic body radiation therapy; Drug: cyclophosphamide; Biological: therapeutic autologous lymphocytes; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: therapeutic autologous lymphocytes — Undergo autologous PBMC infusion
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies the side effects and best way to give stereotactic body radiation therapy and T-cell infusion in treating patients with metastatic kidney cancer. Giving total body irradiation before a T-cell infusion stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and stored. Chemotherapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a safety and feasibility study of stereotactic radiotherapy with autologous T-cell infusion for patients with metastatic renal cell carcinoma.

SECONDARY OBJECTIVES:

I. Determine the progression free survival at one year. II. Determine the overall survival at one year.

OUTLINE:

STEREOTACTIC BODY RADIATION THERAPY (SBRT): Patients undergo standard of care SBRT over 1-2 weeks according to tumor volume and location.

LYMPHODEPLETION: Beginning 3 weeks later, patients receive cyclophosphamide orally (PO) twice daily (BID) for 3 days.

REINFUSION OF PERIPHERAL BLOOD MONONUCLEAR CELLS (PBMC): Within 3-14 days of completing lymphodepletion with cyclophosphamide, patients undergo autologous PBMC infusion.

After completion of study treatment, patients are followed up at 1 week, 4 weeks, and monthly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the kidney (clear-cell predominance)
* Have had at least 2 prior systemic treatments for renal cell carcinoma (RCC)
* Have at least 1 extracranial metastasis that is amenable to radiation and at least 1 other site of disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST)
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Absolute neutrophil count (ANC) >= 0.75 x 10^9/L
* Absolute lymphocyte count (ALC) >= 0.5 X 10^9/L
* Hemoglobin >= 8 g/dL
* Platelets >= 50 X 10^9/L
* Total bilirubin =< 3 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 X ULN
* Serum creatinine =< 2.1 X ULN (or creatinine clearance of > 50 cc/min)

Exclusion Criteria:

* History of other malignancies within 5 years prior to enrollment except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma, squamous-cell carcinoma of the skin, carcinoma in situ of the cervix, early-stage bladder cancer, or low-grade endometrial cancer

  * Malignancies that have undergone a putative surgical cure (i.e., localized prostate cancer post-prostatectomy) within 5 years prior to enrollment may be discussed with the lead primary investigator
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for more than 1 week within 6 months prior enrollment
* Presence of uncontrolled infection
* Evidence of active bleeding or bleeding diathesis; any medical condition requiring systemic anticoagulation (including anti-platelet agents)
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to procedures
* Pregnant and breastfeeding women are excluded; as well as women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control (hormonal or barrier method of birth control; abstinence) to avoid pregnancy for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-related grade 3-5 toxicities, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Within 30 days after infusion of PBMCs
  Adverse events will be tabulated by type and grade at each follow-up interval.

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  The level of OS will be tabulated at each follow-up interval, and will be summarized using Kaplan-Meier curves and medians with 95% confidence intervals.
Progression-free survival (PFS) | The duration from SBRT treatment to documented disease progression or death, assessed at 1 year
  The level of PFS will be tabulated at each follow-up interval. The percentage of individuals free from disease progression will be computed with exact 95% confidence intervals. PFS will be summarized using Kaplan-Meier curves and medians with 95% confidence intervals.

OTHER OUTCOMES:
Level of circulating tumor cells (CTCs) | Up to 2 years
  The correlations of CTCs and changes in signaling as measured by nano-immunoassay (NIA) to clinical response will be assessed. NIA measurements for 20 protein isoforms will be analyzed. Measurements will be analyzed as continuous variables for each sample. The distribution of each isoform will be summarized with medians and interquartile ranges. Quantile plot and box-Cox models will be used to determine whether to transform the data prior to analysis. A protein isoform signature predictive of clinical response will be constructed using the Lasso R glmnet package.
Changes in signaling as measured by NIA | Up to 2 years
  The correlations of CTCs and changes in signaling as measured by NIA to clinical response will be assessed. NIA measurements for 20 protein isoforms will be analyzed. Measurements will be analyzed as continuous variables for each sample. The distribution of each isoform will be summarized with medians and interquartile ranges. Quantile plot and box-Cox models will be used to determine whether to transform the data prior to analysis. A protein isoform signature predictive of clinical response will be constructed using the Lasso R glmnet package.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Srinivas, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States